CLINICAL TRIAL: NCT00617500
Title: Climacteric Clinical Trial : the Use of Complementary Therapy and Hormonal Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sociedade Hospital Samaritano (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Eliseth Ribeiro Leão, Scientific Research Department of Samaritano Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS 18/07
Record Dates: First submitted 2008-01-23; First posted 2008-02-18 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Climacteric
Keywords: climacteric; complementary therapy; hormonal replacement therapy
MeSH Terms: interventions — Therapeutic Touch; Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hormone (Active Comparator)
  Interventions: Drug: Hormones
- flower therapy (Experimental)
  Interventions: Other: flower therapy
- therapeutic touch (Experimental)
  Interventions: Other: therapeutic touch
- auriculotherapy (Experimental)
  Interventions: Other: auricular therapy

INTERVENTIONS:
Other: flower therapy — Each woman will perform 12 sessions of 20 to 30 minutes, depending on the treatment group, with weekly intervals performed in one of the consultation rooms.
  Arms: flower therapy
Other: therapeutic touch — Each woman will perform 12 sessions of 20 to 30 minutes, depending on the treatment group, with weekly intervals performed in one of the consultation rooms.
  Arms: therapeutic touch
Other: auricular therapy — Each woman will perform 12 sessions of 20 to 30 minutes, depending on the treatment group, with weekly intervals performed in one of the consultation rooms.
  Arms: auriculotherapy
Drug: Hormones — Estradiol 1 mg and a drospirenone 2mg/day (3 months)
  Arms: Hormone

SUMMARY:
The alternative and complementary therapies are being gradually included in the Brazilian Health Unique System (SUS), as it is foreseen in the National Politics of Integrative and Complementary Practices in Brazil . However, though this thematic is also included in the National Agenda of Research Priorities concerning Health, published studies concerning this matter are quite scarce. The World Health Organization (WHO) indicated that it is a big challenge to effect the following studies: cost-effectiveness, as well as safety, efficiency and the quality of such practices. WHO also pointed out the clinical situations where they could be applied and that is why this investigation we are undertaken is fully justified.

Annoying signs and symptoms which come along with the climacteric period, especially anxiety, insomnia and hot flushes, change women´s life quality and their affective, social and business relationships as well. Consequently, this can generate sadness, depression and isolation.

Many women cannot undergo hormonal replacement, for several reasons: or they have some illnesses which reject hormones, or due to hypersensitiveness reactions or even economical difficulties. Also, the cost-effectiveness ratio between conventional therapy of hormonal replacement and complementary therapies which compose this study are not known yet .

The complementary therapies proposed in this study concern non-invasive methods, of low cost, which justify being researched in order to verify the potential of those annoying signs alleviation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Recruited and registered in local of the study
* They should present the signs and symptoms checked - insomnia, anxiety and hot flushes, they felt at the beginning of the climacteric
* They should not be under hormonal replacement or even should have stopped their use more than 90 days

Exclusion criteria:

* women who undergo a hysterectomy surgery
* women using hormonal therapy

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 278 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-12 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
annoying signs and climacteric symptoms | pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Study Director — Hospital Samaritano; Maria Julia P Silva, PhD, Study Director — University of Sao Paulo; Léia Sales, MscN, Principal Investigator — University of Sao Paulo; Ivaldo da Silva, PhD, Principal Investigator — Tocogynecological Department of São Paulo Federal University; Maria C Martinez, PhD, Principal Investigator — Hospital Samaritano
Locations (2):
- Brazil (2):
  - Hospital Samaritano, São Paulo, São Paulo
  - Nursing School of University of São Paulo, São Paulo, São Paulo